CLINICAL TRIAL: NCT01382758
Title: Use of Near Infrared Spectroscopy (NIRS) for the Early Detection of Acute Kidney Injury in Children Post Cardiopulmonary Bypass
Brief Title: Near Infrared Spectroscopy for the Detection of Acute Kidney Injury in Children Following Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0527; AAP11-0527 (Other)
Record Dates: First submitted 2011-06-15; First posted 2011-06-27 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-06

CONDITIONS: Acute Kidney Injury; Heart; Dysfunction Postoperative, Cardiac Surgery; Children
Keywords: Near Infrared Spectroscopy (NIRS); Acute kidney injury (AKI)
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Acute kidney injury: The group of patients who develop acute kidney injury as defined by the pediatric RIFLE criteria.
- No acute kidney injury: The patients who do not develop acute kidney injury

SUMMARY:
One in a hundred children is born with a heart defect. Some children require heart surgery within the first few days of life, while others can wait until they are older. A complication of open-heart surgery is low blood flow due to the heart-lung machine that can cause sudden loss of kidney function known as acute kidney injury (AKI). AKI causes complications that can increase hospital length of stay and increase risk of death. Current ways to identify AKI are not able to it until 2 or 3 days after it has occurred. Because of this, there is not a specific treatment for AKI. If the investigators diagnose AKI early, they might be able to treat it and improve outcomes in children. NIRS is a skin monitor that can detect low blood flow to the kidney and might help diagnose AKI when it occurs in the operating room. The use of NIRS to diagnose AKI early is the focus of this study.

DETAILED DESCRIPTION:
Near infrared spectroscopy (NIRS) is a noninvasive tool used for continuous monitoring of regional tissue oxyhemoglobin saturation. Sensors are placed on the head and abdomen or flank and use light to measure the percent oxygen levels in tissues. Head NIRS has been correlated with oxygen levels of the blood returning from the brain, and an abrupt decline in post-operative cardiac patients has been shown in retrospective studies to predict an impending event such as cardiac arrest. Animal studies have demonstrated that somatic NIRS monitoring is able to detect flow-induced changes in regional oxygen levels of the kidney and gut directly under the sensor. Unlike cerebral NIRS monitoring, there is no data regarding the clinical utility of NIRS over the abdomen and flank in predicting outcomes. Children are at risk of decreased organ perfusion following cardiac surgery, and is a phenomenon termed low cardiac output syndrome (LCOS). It occurs in approximately 25% of neonates and young children following cardiac surgery. The effects of LCOS on end organ function, specifically the kidney may result in acute kidney injury, thereby increasing morbidity and mortality. The incidence of acute kidney injury (AKI) following cardiac surgery is reported as high as 40%. The use of NIRS in the operating room to detect AKI in pediatric patients undergoing cardiac surgery is the focus of this proposal Specific Aim 1: Determine if a reduction in renal NIRS intra-operatively identifies patients with AKI Hypothesis: Reduced intra-operative renal NIRS will precede the diagnosis of acute kidney injury by an increase in serum creatinine within 1 to 3 days post-cardiopulmonary bypass Specific Aim 2: Determine if a reduction in renal NIRS intra-operatively correlates with increases in emerging biomarkers of AKI.

Hypothesis: Reduced intra-operative renal NIRS will precede the development if AKI as detected by neutrophil gelatinase-associated lipocalin, IL-6 and IL-18 by at least 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* All children less than or equal to age 4 undergoing cardiac surgery with the use of cardiopulmonary bypass at Colorado Children's Hospital

Exclusion Criteria:

* Prior enrollment in the study
* Agre greater than 4 years
* Use of nephrotoxic drugs within 48 hours of surgery
* Underlying renal dysfunction (preoperative estimated Schwartz clearance less than 80ml/min/1.73m2)
* Gestational age less than 34 weeks at the time of surgery
* Withdrawal of care planned

Ages: 1 Day to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children undergoing cardiac surgery with the use of cardiopulmonary bypass at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 48-72 hours
  A decline in intra-operative renal NIRS to predict AKI as measured by an increase in serum creatinine. Baseline lab testing, including BMP, UA. Renal NIRS sensors will be placed prior surgery. In the OR, continuous real time monitoring of NIRS will occur and continue for 72 hours after cardiopulmonary bypass (CPB). BMP will be performed after surgery and at 24, 48 and 72 hours. Repeat UA will be performed at 24 hours post CPB, and urine electrolytes and urea will be performed at 12, 24, 48 and 72 hours. AKI as defined by the pRIFLE criteria at 48-72 hours post cardiopulmonary bypass.

SECONDARY OUTCOMES:
Acute kidney injury by renal biomarkers | 12 hours
  NIRS monitoring as described above. Baseline renal biomarkers (urine: NGAL, IL-18, IL-6, serum: IL-6, IL-8) followed by repeated sampling at 6, 12, 24, 48 and 72 hours post initiation of CPB. Serum sampling will last only occur through 24 hours.
Mechanical ventilation and acute kidney injury | Hospital admission (day 1)
  Duration of mechanical ventilation, including any failures of extubation. Will include ventilator parameters (inspired oxygen, peak pressures)
Hospital length of stay and AKI | An average of 1 week for simple defects and 4 weeks for complex congenital heart defects (Hypoplastic left heart syndrome)
  Evaluate intensive care and hospital length of stay with regards to presence or absence of AKI
30-day mortality and AKI | 30 days
  Evaluate the 30-day mortality with regards to presence or absence of AKI

CONTACTS AND LOCATIONS:
Overall Officials: Katja Gist, DO, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Background] Wider M. Monitoring regional hemoglobin oxygen saturation (rSO2) of the kidney and gut. Somanetics corporation
- [Background] Hoffman GM, Stuth EA, Jaquiss RD, Vanderwal PL, Staudt SR, Troshynski TJ, Ghanayem NS, Tweddell JS. Changes in cerebral and somatic oxygenation during stage 1 palliation of hypoplastic left heart syndrome using continuous regional cerebral perfusion. J Thorac Cardiovasc Surg. 2004 Jan;127(1):223-33. doi: 10.1016/j.jtcvs.2003.08.021. PMID 14752434
- [Background] Kaufman J, Almodovar MC, Zuk J, Friesen RH. Correlation of abdominal site near-infrared spectroscopy with gastric tonometry in infants following surgery for congenital heart disease. Pediatr Crit Care Med. 2008 Jan;9(1):62-8. doi: 10.1097/01.PCC.0000298640.47574.DA. PMID 18477915
- [Background] Kussman BD, Wypij D, Laussen PC, Soul JS, Bellinger DC, DiNardo JA, Robertson R, Pigula FA, Jonas RA, Newburger JW. Relationship of intraoperative cerebral oxygen saturation to neurodevelopmental outcome and brain magnetic resonance imaging at 1 year of age in infants undergoing biventricular repair. Circulation. 2010 Jul 20;122(3):245-54. doi: 10.1161/CIRCULATIONAHA.109.902338. Epub 2010 Jul 6. PMID 20606124
- [Background] Mishra J, Dent C, Tarabishi R, Mitsnefes MM, Ma Q, Kelly C, Ruff SM, Zahedi K, Shao M, Bean J, Mori K, Barasch J, Devarajan P. Neutrophil gelatinase-associated lipocalin (NGAL) as a biomarker for acute renal injury after cardiac surgery. Lancet. 2005 Apr 2-8;365(9466):1231-8. doi: 10.1016/S0140-6736(05)74811-X. PMID 15811456
- [Background] Parikh CR, Mishra J, Thiessen-Philbrook H, Dursun B, Ma Q, Kelly C, Dent C, Devarajan P, Edelstein CL. Urinary IL-18 is an early predictive biomarker of acute kidney injury after cardiac surgery. Kidney Int. 2006 Jul;70(1):199-203. doi: 10.1038/sj.ki.5001527. Epub 2006 May 17. PMID 16710348
- [Background] Akcan-Arikan A, Zappitelli M, Loftis LL, Washburn KK, Jefferson LS, Goldstein SL. Modified RIFLE criteria in critically ill children with acute kidney injury. Kidney Int. 2007 May;71(10):1028-35. doi: 10.1038/sj.ki.5002231. Epub 2007 Mar 28. PMID 17396113
- [Background] Ferrari M, Mottola L, Quaresima V. Principles, techniques, and limitations of near infrared spectroscopy. Can J Appl Physiol. 2004 Aug;29(4):463-87. doi: 10.1139/h04-031. PMID 15328595
- [Background] Dent CL, Ma Q, Dastrala S, Bennett M, Mitsnefes MM, Barasch J, Devarajan P. Plasma neutrophil gelatinase-associated lipocalin predicts acute kidney injury, morbidity and mortality after pediatric cardiac surgery: a prospective uncontrolled cohort study. Crit Care. 2007;11(6):R127. doi: 10.1186/cc6192. PMID 18070344
- [Background] Liu KD, Altmann C, Smits G, Krawczeski CD, Edelstein CL, Devarajan P, Faubel S. Serum interleukin-6 and interleukin-8 are early biomarkers of acute kidney injury and predict prolonged mechanical ventilation in children undergoing cardiac surgery: a case-control study. Crit Care. 2009;13(4):R104. doi: 10.1186/cc7940. Epub 2009 Jul 1. PMID 19570208
- [Background] Dennen P, Altmann C, Kaufman J, Klein CL, Andres-Hernando A, Ahuja NH, Edelstein CL, Cadnapaphornchai MA, Keniston A, Faubel S. Urine interleukin-6 is an early biomarker of acute kidney injury in children undergoing cardiac surgery. Crit Care. 2010;14(5):R181. doi: 10.1186/cc9289. Epub 2010 Oct 13. PMID 20942931
- [Background] Kist-van Holthe tot Echten JE, Goedvolk CA, Doornaar MB, van der Vorst MM, Bosman-Vermeeren JM, Brand R, van der Heijden AJ, Schoof PH, Hazekamp MG. Acute renal insufficiency and renal replacement therapy after pediatric cardiopulmonary bypass surgery. Pediatr Cardiol. 2001 Jul-Aug;22(4):321-6. doi: 10.1007/s002460010238. PMID 11455401
- [Background] Bennett M, Dent CL, Ma Q, Dastrala S, Grenier F, Workman R, Syed H, Ali S, Barasch J, Devarajan P. Urine NGAL predicts severity of acute kidney injury after cardiac surgery: a prospective study. Clin J Am Soc Nephrol. 2008 May;3(3):665-73. doi: 10.2215/CJN.04010907. Epub 2008 Mar 12. PMID 18337554